CLINICAL TRIAL: NCT07022366
Title: Investigating the Neuropsychological Effects of 5-HT2a Antagonism
Acronym: PANDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R95550/RE001
Record Dates: First submitted 2025-05-27; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: serotonin 2a; pimavanserin
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pimavanserin (Experimental): Single dose of pimavanserin (10mg)
  Interventions: Drug: Pimavanserin 10mg
- Placebo (Placebo Comparator): Single dose of matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin 10mg — Single dose of pimavanserin (10mg)
  Arms: Pimavanserin
Drug: Placebo — Sucrose tablet
  Arms: Placebo

SUMMARY:
Serotonin is an important chemical in the brain that helps control mood, sleep, and appetite. Most antidepressant medications work by affecting serotonin to help improve symptoms. A serotonin receptor is like a "lock" on the surface of brain cells, and serotonin acts like a "key" that fits into these locks. When serotonin binds to the receptor, it sends a signal that helps control different functions in the brain, like mood and behavior. There are different types of serotonin receptors, and each one affects different parts of the brain. Pimavanserin is a medication licensed in the United States of America for the treatment of patients with Parkinson's Disease. It has a very specific effect on one type of serotonin receptor (the serotonin 2a receptor). In this study, the investigators will use pimavanserin to understand more about this serotonin receptor, which may help develop new treatments for depression in the future. More specifically, the study will focus on how pimavanserin impacts cognitive functions such as memory, how we process emotional information and how we make decisions, and will compare these effects to a placebo (a treatment that doesn't have active ingredients).

DETAILED DESCRIPTION:
Serotonin (5-HT) 2A receptors are widely expressed in the human brain in areas involved in cognition and emotion and are thought to play a key role in the aetiology of a number of psychiatric disorders, including depression. Medication free patients with depression have increased 5-HT2A receptor binding (Bhagwagar et al., 2006) and many effective antidepressant treatments are antagonists of the 5-HT2A receptor, including mirtazapine, olanzapine, quetiapine and aripiprazole. Conversely, psychedelic drugs such as psilocybin are powerful agonists of the 5-HT2A receptor, and are gaining traction as a novel approach to the treatment of depression (Goodwin et al 2022).

Animal and human studies suggest that the 5-HT2A receptor plays a key role in memory and cognitive flexibility. Activation of the 5-HT2A receptor in animals has been shown to improve novel object memory, with a particular effect on the consolidation of memories (Zhang et al 2012). There is also an increasing body of evidence suggesting that 5-HT2A agonists may increase cognitive flexibility, and this is thought to be one mechanism through which psychedelics may exert their rapid-onset and sustained antidepressant effects (Luppi et al 2024). For example, the non-selective 5-HT2A receptor agonist lysergic acid diethylamide (LSD) has been shown to increase learning rates and exploratory behaviour on a probabilistic reversal learning task in healthy volunteers (Kanen et al 2022), which is consistent with increased flexibility and a destabilisation of existing beliefs/priors.

However, the existing evidence base is somewhat mixed, with contradictory findings regarding the direction of effects of 5-HT2A activation on cognition. It is likely that this is in part due to the non-selective nature of the pharmacological probes used, with many having effects on serotonin receptors beyond 5-HT2A and on other neurotransmitter systems, including dopamine. There is also evidence that 5-HT2A agonists that have psychedelic properties may have a unique profile of effects on intracellular 5-HT2A receptors (Vargas et al 2023), which further complicates the interpretation of the existing evidence base.

The development of highly selective 5-HT2A antagonists offers the opportunity to further understand the role played by this receptor subtype in cognition. Pimavanserin has a relatively selective pharmacological action; it is a potent inverse agonist of the 5-HT2A receptor and also has around 40-fold less potent activity at 5-HT2C receptors. Pimavanserin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of hallucinations and delusions associated with psychosis in people with Parkinson's disease with a recommended dose range between 34-40mg once daily. Whilst at this dose it is likely that both 5-HT2A and 5-HT2C receptors are engaged, Positron Emission Tomography (PET) studies have demonstrated that with lower doses (10-20mg) it is possible to achieve full saturation of the 5-HT2A receptor without action at the 5-HT2C receptor (Nordstrom et al 2007). The effects of pimavaserin have also been tested in patients with depression in a study in which it was administered as an adjunct to standard antidepressant treatment. Whilst there were some initial positive findings of benefits on depressive symptoms, impulsivity, irritability, anxiety, insomnia, daytime sleepiness, and sexual and psychosocial functioning (Fava et al 2019), subsequent Phase 3 trials were less positive (Dirks et al 2022). Pimavanserin is well tolerated with minimal side effects; the most common side effects reported in the trials were dry mouth, nausea and headache. Low dose pimavanserin therefore offers the opportunity to safely and selectively manipulate the function of 5-HT2A receptors in the human brain.

In this study, the investigators will use pimavanserin as a pharmacological probe to further investigate the role of the 5-HT2A receptor in human cognition. Healthy volunteers will be randomised to receive a single dose (10mg) of pimavanserin or placebo. Four hours later (once the drug has reached peak plasma concentration), they will complete a battery of cognitive tests designed to measure learning and memory, cognitive flexibility and emotional processing. The investigators will also collect sleep monitoring data from a sub-set of participants for a feasibility study. The monitoring of sleep is a useful metric to consider as it may uncover further details pimavanserin's mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the research
* Aged 18-45 years
* Good vision and hearing
* Body mass index (BMI) within the range of 18-35kg/m2 (This is to ensure an appropriate pharmacokinetic profile for pimavanserin is achieved by all participants)
* Sufficiently fluent in English to understand tasks
* Willing to avoid drinking any alcohol the day before the research visit

Exclusion Criteria:

* Currently receiving or seeking treatment for any mental health condition
* Any past or current history of severe and/or serious psychiatric disorder, including but not limited to schizophrenia, psychosis, bipolar affective disorder, severe major depressive disorder, obsessive compulsive disorder (covered in SCID-5 assessment in screening procedures)
* ADHD requiring treatment with stimulant or other centrally-acting drugs
* Regular alcohol consumption of more than 21 units per week
* A head injury causing concussion or unconsciousness in the past 6 months
* Pregnancy / intention to become pregnant during the study or breastfeeding
* Any use of recreational drugs in the last three months
* Participation in any other drug study in the last three months
* Participation in any other study with the same tasks in the last year
* History of cardiac disease or cardiac arrhythmias
* Prolonged QTc interval on baseline ECG
* Current usage of other drugs known to prolong QT interval including Class 1A or 3 antiarrhythmics, e.g. certain antibiotics (getifloxacin, moxifloxacin)
* Current use of drugs that inhibit CYP3A4 (eg Clarithromycin. Diltiazem. Erythromycin. Fluconazole). Participants will be asked to avoid grapefruit juice in the week before the study.
* Current use of psychoactive medication that in the opinion of the Chief Investigator may interfere with the study measures
* History of, or current medical condition(s) which, in the opinion of the Investigator may interfere with the safety of the participant or the scientific integrity of the study, including epilepsy/seizures, brain injury, severe hepatic or renal disease, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, severe neurological problems (e.g. Parkinson's disease; blackouts requiring hospitalisation);
* Any physical (including visual and auditory), cognitive or language impairment that would make complying with the study protocol challenging
* Excessive caffeine consumption, i.e., consumption higher than 8 cups of standard caffeinated drinks (tea, instant coffee) or higher than 6 cups of stronger coffee or other drinks containing methylxanthines such as coca cola or Red Bull per day;
* Smoking >10 cigarettes per day; or equivalent nicotine consumption
* Participant who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the chief investigator.
* Inability to ingest up to 95mg of lactose

Additional Exclusion Criteria for Participants in the Sleep Study Cohort:

* Unable to undergo cardiac monitoring
* Unable to wear the sleep patch device for full monitoring period
* Implanted neurostimulator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity to loss and reward | 6-8 hours post-intervention
  Choice behaviour on the Probabilistic Reversal Learning Task (PRL)

SECONDARY OUTCOMES:
Emotional memory | 6-8 hours post-intervention
  Performance (accuracy and reaction time) on emotional encoding and recall/recognition memory tasks
Facial expression recognition | 6-8 hours post-intervention
  Performance (accuracy, reaction time and misclassifications) on Facial Expression Recognition Task (FERT
Behavioural response inhibition | 6-8 hours post-intervention
  Performance (accuracy/response time) on Emotional Go/No-Go (EGNG) task
Cognitive Flexibility | 6-8 hours post-intervention
  Performance on the Probabilistic Reversal Learning and the Wisconsin Card Sorting Task
Sleep | Night following pimavanserin administration
  Cardiorespiratory parameters from chest electrocardiogram (ECG) and impedance pneumography (IP) patches, including total sleep time and time in light (N1-2), deep (N3) and REM sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Vargas MV, Dunlap LE, Dong C, Carter SJ, Tombari RJ, Jami SA, Cameron LP, Patel SD, Hennessey JJ, Saeger HN, McCorvy JD, Gray JA, Tian L, Olson DE. Psychedelics promote neuroplasticity through the activation of intracellular 5-HT2A receptors. Science. 2023 Feb 17;379(6633):700-706. doi: 10.1126/science.adf0435. Epub 2023 Feb 16. PMID 36795823
- [Background] Nordstrom AL, Mansson M, Jovanovic H, Karlsson P, Halldin C, Farde L, Vanover KE, Hacksell U, Brann MR, Davis RE, Weiner DM. PET analysis of the 5-HT2A receptor inverse agonist ACP-103 in human brain. Int J Neuropsychopharmacol. 2008 Mar;11(2):163-71. doi: 10.1017/S1461145707007869. Epub 2007 Aug 21. PMID 17708779
- [Background] Luppi AI, Girn M, Rosas FE, Timmermann C, Roseman L, Erritzoe D, Nutt DJ, Stamatakis EA, Spreng RN, Xing L, Huttner WB, Carhart-Harris RL. A role for the serotonin 2A receptor in the expansion and functioning of human transmodal cortex. Brain. 2024 Jan 4;147(1):56-80. doi: 10.1093/brain/awad311. PMID 37703310
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843
- [Background] Dirks B, Fava M, Atkinson SD, Joyce M, Thase ME, Howell B, Lin T, Stankovic S. Adjunctive Pimavanserin in Patients with Major Depressive Disorder: Combined Results from Two Randomized, Double-Blind, Placebo-Controlled Phase 3 Studies. Psychopharmacol Bull. 2022 Oct 27;52(4):8-30. doi: 10.64719/pb.4448. PMID 36339271
- [Background] Bhagwagar Z, Hinz R, Taylor M, Fancy S, Cowen P, Grasby P. Increased 5-HT(2A) receptor binding in euthymic, medication-free patients recovered from depression: a positron emission study with [(11)C]MDL 100,907. Am J Psychiatry. 2006 Sep;163(9):1580-7. doi: 10.1176/ajp.2006.163.9.1580. PMID 16946184